CLINICAL TRIAL: NCT01157260
Title: The Effects of AST-120 on Endothelial Dysfunction in Patients With Chronic Kidney Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ewha Womans University (Other)
Responsible Party: Nephrology, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ewha AST-120
Record Dates: First submitted 2010-06-25; First posted 2010-07-07 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-03

CONDITIONS: Kidney Failure, Chronic
Keywords: Indoxyl sulfate; AST-120
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — AST 120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AST-120 (Experimental): AST-120 administration 2g three times a day
  Interventions: Drug: Kremezin
- Control (No Intervention): Control Chronic Kidney disease stage 3,4

INTERVENTIONS:
Drug: Kremezin — AST-120 2g three times a day
  Other Names: AST-120 (Kremezin) 2g three times a day
  Arms: AST-120

SUMMARY:
Indoxyl sulfate (IS) is a uremic toxin that accelerates the progression of chronic kidney disease (CKD). AST-120 (Kremezin®; Kureha Corporation, Tokyo, Japan) removes indole, which is the precursor of IS, in the intestine, and reduces the accumulation of IS. This drug has been shown to retard the deterioration of renal function in CKD patients through reducing the levels of IS.

IS was reported to promote aortic calcification and stimulate the proliferation of vascular smooth muscle cells (VSMC). IS also inhibits endothelial proliferation and wound repair. With this background, the investigators will performed the study whether AST-120 improve the endothelial dysfunction in CKD patients.

DETAILED DESCRIPTION:
The purpose of this study is to examine whether Kremezin, Indoxyl sulfate lowering agent improve endothelial dysfunction in stage 3,4 chronic kidney disease patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic kidney disease (Stage3 - Stage4)
* Patients who are able and willing to understand, sign and date an informed consent document, and authorize access to protected health information

Exclusion Criteria:

* Acute gastric or duodenal ulcer
* Severe constipation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Changes of FMD(Flow Mediated Dilatation) | 6 months
  FMD (Flow Mediated Dilatation): percent change of FMD response to hyperemia and after sublingual nitroglycerin on brachial artery.

SECONDARY OUTCOMES:
Level of Indoxyl Sulfate | 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hee Kang, MD. PhD., Principal Investigator — Ewha Womans University
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea